CLINICAL TRIAL: NCT03730207
Title: A Prospective, 1: 1 Randomized, Single Blind, Multi-center Human Clinical Trial
Brief Title: Xpede Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDT17075SD1707
Record Dates: First submitted 2018-10-16; First posted 2018-11-05 (Actual); Results first posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Pathological Fracture of Vertebra Due to Secondary Osteoporosis (Disorder); Pathological Fracture of Vertebra Due to Neoplastic Disease (Disorder)

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Xpede™ Bone Cement (Experimental): The subjects in this group will be injected the Xpede™ Bone Cement into vertebral body via percutaneous Vertebroplasty or Kyphoplasty to stabilize the fractured vertebral body.
  Interventions: Device: Xpede™ Bone Cement
- Mendec Spine Bone Cement (Active Comparator): The subjects in this group will be injected the Mendec Spine Bone Cement into vertebral body via percutaneous Vertebroplasty or Kyphoplasty to stabilize the fractured vertebral body.
  Interventions: Device: Mendec Spine Bone Cement

INTERVENTIONS:
Device: Xpede™ Bone Cement — Xpede™ Bone Cement will be injected into vertebral body via percutaneous Vertebroplasty or Kyphoplasty to stabilize the fractured vertebral body by filling the bony trabeculae.
  Arms: Xpede™ Bone Cement
Device: Mendec Spine Bone Cement — Mendec Spine Bone Cement will be injected into vertebral body via percutaneous Vertebroplasty or Kyphoplasty to stabilize the fractured vertebral body by filling the bony trabeculae.
  Arms: Mendec Spine Bone Cement

SUMMARY:
The purpose of this clinical study is to confirm the efficacy and safety of the Kyphon®Xpede™ Bone Cement in human use in China.

ELIGIBILITY:
Inclusion Criteria:

1. Subject being diagnosed as having painful pathological vertebral body fracture, who is suitable for VP/BKP procedure (1-3 levels) according to clinic practice.
2. Subjects who are willing to participate in study through consent and willing to undergo study specific required procedures with expectancy of geographically stable for follow up duration.
3. Subjects are at least 18 and ≤80 years old .

Exclusion Criteria:

1. Subject has a local or systemic infection.
2. Subject has pains caused by other spine disease than painful pathological vertebral compression fracture.
3. Subject has a medical condition with less than 1 year of life expectancy.
4. Subject is grossly obese, i.e. BMI≥40.
5. Subject has medical conditions that represent contraindications for the use of bone cement by investigator's decision.
6. Subject has an allergy or an intolerance to bone cement component.
7. Subject has past spinal surgeries at the target level(s) for which the VP/BKP procedure is suitable.
8. Subjects who are currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent trials is only allowed when document pre-approval is obtained from the Medtronic study manager and Medtronic Medical Advisor.
9. Pregnant women or breastfeeding women, or women of child bearing potential who are not on a reliable form of birth regulation method or abstinence.
10. Subjects with exclusion criteria required by local law (age or other).
11. Subjects with medical condition which precludes them from participation in the opinion of the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan
  - Hunan provincial people's hospital, Changsha, Hunan
  - The first affiliated hospital of Suzhou university, Suzhou, Jiangsu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Started | 89 | 91
Completed | 83 | 88
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement | Total
Number analyzed (Participants) | 89 | 91 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (5.59) | 67.1 (7.06) | 67.6 (6.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 89 | 91 | 180
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 89 | 91 | 180

OUTCOME MEASURES:

1. Primary Outcome: The Change of Numerical Rating Scale (NRS) Score From Baseline at 6 Months Postoperative
Description: NRS is used for rating patient pain intensity from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be."
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 83 | 88
score | -4.2 (2.86) | -4.4 (2.76)

2. Primary Outcome: The Change of Index Vertebral Body Angle From Baseline at 6 Months
Description: Vertebral body angle is defined the angle formed by lines drawn parallel to the superior endplate of the fractured vertebral body and the inferior endplate of the fractured vertebral body for each fractured vertebral body.
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: degree
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 71 | 79
degree | -0.869 [-1.817 to 0.078] | -0.952 [-1.878 to -0.027]

3. Secondary Outcome: The Change of NRS Score From Baseline at 1 Day and 3 Months
Description: as for outcome 1
Time Frame: Baseline, 1 day, and 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 89 | 91
score
  The change of NRS score from baseline at 1 day | -2.9 [-3.5 to -2.3] | -2.3 [-2.9 to -1.7]
  The change of NRS score from baseline at 3 months | -3.6 [-4.2 to -3.1] | -3.8 [-4.4 to -3.3]

4. Secondary Outcome: The Change of Oswestry Disability Index (ODI) Score From Baseline at 1 Day, 3 Months, and 6 Months
Description: ODI Questionnaire is used to assess patient back function. The ODI score ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
Time Frame: Baseline, 1 day, 3 months, and 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 89 | 91
score on a scale
  The change of ODI score from baseline 3 months | -26.407 [-31.714 to -21.100] | -29.108 [-34.331 to -23.885]
  The change of ODI score from baseline 6 months | -26.407 [-31.714 to -21.100] | -29.108 [-34.331 to -23.885]
  The change of ODI score from baseline 1 day | -1.757 [-7.297 to 3.782] | 1.746 [-3.698 to 7.190]

5. Secondary Outcome: The Change of SF-36 From Baseline at 1 Day, 3 Months, and 6 Months
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) is used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS/MCS is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: Baseline, 1 day, 3 months, and 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 89 | 91
score on a scale
  The change of SF-36(MCS)from baseline at 6 months | 3.781 [-0.106 to 7.668] | -1.436 [-5.190 to 2.317]
  The change of SF-36(MCS) from baseline at 3 months | 5.740 [2.018 to 9.462] | 0.086 [-3.498 to 3.671]
  The change of SF-36(MCS)from baseline at 1 day | 0.650 [-2.591 to 3.890] | 0.809 [-2.293 to 3.911]
  The change of SF-36(PCS)from baseline at 6 months | 7.855 [4.838 to 10.872] | 9.683 [6.725 to 12.641]
  The change of SF-36(PCS)from baseline at 3 months | 5.740 [2.783 to 8.697] | 6.504 [3.605 to 9.404]
  The change of SF-36(PCS)from baseline at 1 day | -3.104 [-5.596 to -0.611] | -3.654 [-6.097 to -1.211]

6. Secondary Outcome: Change in Vertebral Body Height at 1 Day, 3 Months, and 6 Months
Description: Vertebral Body Height in the lateral projection will be measured at each treated vertebra as well as the next adjacent vertebrae (superior and inferior) without fracture and reported in millimeters.
  Vertebral Body Height is the distance between comparable points on the superior and inferior endplates of the vertebral body at the posterior (Hp), midline (Hm) and anterior (Ha) locations。
Time Frame: 1 day, 3 months, and 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: millimetre
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 89 | 91
millimetre
  Change in vertebral body height (Anterior height) restoration at 6 months | -4.271 [-5.348 to -3.195] | -4.429 [-5.492 to -3.366]
  Change in vertebral body height (Anterior height) restoration at 3 months | -3.949 [-5.040 to -2.859] | -4.154 [-5.234 to -3.074]
  Change in vertebral body height (Anterior height) restoration at 1 day | -2.514 [-3.597 to -1.432] | -2.738 [-3.809 to -1.666]
  Change in vertebral body height (Mid-vertebral height) restoration at 1 day | -2.375 [-2.375 to -1.531] | -2.845 [-3.679 to -2.011]
  Change in vertebral body height (Mid-vertebral height) restoration at 3 months | -3.727 [-4.610 to -2.844] | -3.979 [-4.850 to -3.108]
  Change in vertebral body height (Mid-vertebral height) restoration at 6 months | -3.426 [-4.255 to -2.597] | -3.603 [-4.418 to -2.788]
  Change in vertebral body height (Posterior height) restoration at 1 day | -0.128 [-0.912 to 0.656] | -0.613 [-1.387 to 0.160]
  Change in vertebral body height (Posterior height) restoration at 3 months | -0.821 [-1.682 to 0.041] | -1.579 [-2.426 to -0.732]
  Change in vertebral body height (Posterior height) restoration at 6 months | -0.862 [-1.628 to -0.096] | -1.451 [-2.201 to -0.702]

7. Secondary Outcome: Change in Vertebral Body Angle From Baseline at 1 Day and 3 Months
Description: as for outcome 2
Time Frame: Baseline, 1 day and 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: degree
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 86 | 90
degree
  Change in Vertebral body angle from baseline at 3 months | -1.710 [-2.693 to -0.727] | -1.662 [-2.629 to -0.695]
  Change in Vertebral body angle from baseline at 1 day | -2.739 [-3.629 to -1.848] | -2.375 [-3.254 to -1.496]

8. Secondary Outcome: Number of Participants With Adverse Events Reported Through 6 Months
Description: Adverse events reported through 6 months, in particular, the following events will be reported:
  * Bone Cement Implantation Syndrome;
  * Bone Cement leakage;
  * Vertebral body compression fracture;
  * Adjacent vertebral body fracture;
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
Number analyzed (Participants) | 89 | 91
Participants | 28 | 32

ADVERSE EVENTS:
Time Frame: The mean (±sd) total duration of study exposure was 196.3±49.49 days.
Arm/Group | Xpede™ Bone Cement | Mendec Spine Bone Cement
All-Cause Mortality (participants affected / at risk) | 2/89 | 1/91
Serious Adverse Events (participants affected / at risk) | 1/89 | 1/91
Other Adverse Events (participants affected / at risk) | 12/89 | 7/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Xpede™ Bone Cement (N=89) | Mendec Spine Bone Cement (N=91)
Multiple organ failure (General disorders) | 1 (1) | 0 (0)
Post-operative recurrence of right breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/32 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xpede™ Bone Cement (N=89) | Mendec Spine Bone Cement (N=91)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 12 (12) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT03730207/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT03730207/SAP_001.pdf